CLINICAL TRIAL: NCT05300659
Title: Feasibility of an Upper Limb Functional Training Programme to Support Self-management in Stroke Survivors (ASTAR)
Brief Title: A STudy of Upper Arm Rehabilitation in Stroke Survivors- ASTAR
Acronym: ASTAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Khalid Ali (Other)
Collaborators: ARNI Institute for Neurological Rehabilitation (ARNI) (Unknown)
Responsible Party: Sponsor-Investigator, Dr Khalid Ali, Senior lecturer in Geriatrics, BSMS, Brighton & Sussex Medical School
Organization: Brighton & Sussex Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRAS-254799
Record Dates: First submitted 2022-03-16; First posted 2022-03-29 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Stroke; Upper Limb Injury; Rehabilitation
MeSH Terms: conditions — Stroke; Arm Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Blinded research nurse will take upper limb measurements at baseline, after 10 therapy sessions and at 6 months follow up, without knowing which of the two groups participant had been randomized to .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention)
- ARNI care (Experimental)
  Interventions: Other: Action for Rehabilitation for Neurological Injury (ARNI)

INTERVENTIONS:
Other: Action for Rehabilitation for Neurological Injury (ARNI) — If randomised to upper limb training, a patient will undertake 10 therapy sessions with an instructor from the Action for Rehabilitation for Neurological Injury (ARNI) program during their hospital stay. The last two ARNI-led sessions will be filmed by a nurse/carer on either their own tablet/phone or an i-pad. Participants in the ARNI group will be encouraged to continue doing their personalized exercises while in hospital and continued at home. They will also be given a task-training board to take home
  Arms: ARNI care

SUMMARY:
This feasibility study will explore the clinical effectiveness of additional upper limb therapy compared to standard care delivered to Stroke Survivors at Sussex Rehabilitation Centre (SRC). Randomization via sealed envelope will allocate treatment group to either routine care or upper limb training for self-management plus routine care. If randomized to upper limb training, a patient will undertake 10 therapy sessions with an instructor from the Action for Rehabilitation for Neurological Injury (ARNI) program during their hospital stay. The last two ARNI-led sessions will be filmed by a nurse/carer on either their own tablet/phone or an i-pad. Participants in the ARNI group will be encouraged to continue doing their personalized exercises while in hospital and continued at home. The participants in the ARNI group will also be given a task-training board to take home.

This randomized controlled trial will measure outcomes of each group over six months. Each patient in the study will have upper limb physical measurements taken by a blinded Research Nurse (RN2) at baseline. Research Nurse (RN1) will gather data in a Clinical Report File from a weekly exercise diary completed by the patient or carer and well-being questionnaires. On discharge, RN2 will conduct upper limb measurements, collect completed hospital diaries and issue new ones to take4 home. RN1 will give a weekly phone call or text reminders so that patients to complete exercise diaries at home. At 6 months RN2 will do final measurements and complete patient questionnaires in an out patients clinic visit.

The investigators aim to recruit 36 patients and anticipate 30(8.3%) will complete the 6 month follow-up.

The study sponsor will be the University of Sussex. However, as the study is run in rehabilitation unit in an NHS hospital, University Hospitals Sussex NHS Trust will host the study.

ELIGIBILITY:
Inclusion Criteria:

* Stroke Survivors admitted to Sussex Rehabilitation Centre
* Aged 18 years or over
* Have an upper limb affected by stroke
* Have capacity to consent to participate in the study
* Medically stable

Exclusion Criteria:

* Aged under 18 years
* AMTS <8
* Have a neurological deficit which does not involve upper limb
* Presence of a terminal illness with shortened life expectancy <6 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-07-08 (Estimated); Study Completion 2023-07-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants retained in this feasibility study. | 6 months
  Investigators hypothesize that an ARNI approach to upper limb therapy following stroke will be feasible to implement in a standard NHS rehabilitation unit resulting in better upper limb recovery through providing more intensity and enhancing self-management. If the study proves to be feasible - retention of at least 30/36 patients and at least 70% of data relating to exercise intensity, it can be rolled out to several rehabilitation units across the UK. A follow-up multi-centre randomized controlled trial of ARNI-led upper limb therapy plus usual care compared to usual care will then be carried out to provide clinical and cost effectiveness of the ARNI approach. Upper limb function outcomes: Fugl-Meyer test, Action Research Arm Test. Some questionnaires will be used to assess the psychological well-being of patients and carers: Stroke self-efficacy questionnaire, Stroke carer burden scale (CBS), Stroke specific QOL scale, Stroke Impact Scale (SIS) and EQ-5D.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Sussex NHS Foundation Trust - Sussex Rehabilitation Centre, Haywards Heath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
By request to the Chief Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 3years of study commencement